CLINICAL TRIAL: NCT05033938
Title: Patient Satisfaction With Early Wrist Mobilization Following Volar Locking Plate Fixation of Distal Radius Fractures - a Prospective Randomized Clinical Trial
Brief Title: Early Mobilization Following Volar Locking Plate Fixation of Distal Radius Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert Wood Johnson Barnabas Health (Other)
Collaborators: Brielle Orthopedics (Unknown); Universtiy Orthopedics Associates (Unknown)
Responsible Party: Principal Investigator, Bobby Varghese, MD, Research Assistant, Robert Wood Johnson Barnabas Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mod2021000381
Record Dates: First submitted 2021-07-22; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Distal Radius Fracture
Keywords: volar locking plate; wrist fracture; plates and screws
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Mobilization (Active Comparator): Post-operatively subjects receive a removable wrist splint that can be taken off for early wrist mobilization
  Interventions: Procedure: Early Mobilization Protocol
- Late Mobilization (Active Comparator): Post-operatively subjects receive a splint and are not instructed to not move their wrist till the 2 week follow up visit.
  Interventions: Procedure: Late Mobilization Protocol

INTERVENTIONS:
Procedure: Early Mobilization Protocol — Subjects will be placed in a bulky soft dressing immediately after surgery. They will be made non-weight bearing, but active and passive motion of digits, forearm, elbow, and shoulder will be allowed with light functional tasks permitted as tolerated. Wrist motion within the soft dressing will be permitted as tolerated by patient. On postoperative day 3, patients will be advised to remove the dressing at home and begin home hand/wrist therapy. They will use a removable Velcro wrist splint for nighttime wear and strenuous activity. This splint can be removed during normal activities of daily living and therapy.
  Arms: Early Mobilization
Procedure: Late Mobilization Protocol — Subjects will be placed in a plaster volar resting splint. They will be made non-weight bearing, with use of digits for light functional tasks permitted. They will be given home exercises for their fingers but will not yet resume wrist motion
  Arms: Late Mobilization

SUMMARY:
The overall purpose of this study is to establish the utility of early mobilization in improving patient satisfaction following plate and screw fixation of wrist fractures. Subjects will have objective range of motion data collected and subjective survey data collected at 2 weeks, 6 weeks, 3 months, and 1 year after being randomized either to an early mobilization group that receives a removable wrist splint or a late mobilization group that is placed in a splint for 2 weeks post-operatively. The investigators expect that early wrist mobilization following locking plate fixation of wrist fractures will lead to an increase in postoperative patient satisfaction without a significant increase in complications.

DETAILED DESCRIPTION:
This study will be a prospective randomized clinical trial which will explore differences in outcomes between early and late mobilization in patients undergoing volar plate fixation of distal radius fractures (DRF). The data will be collected at two weeks, six weeks, three months, and one year postoperatively. Data will be collected utilizing questionnaires, in-office measurements, and radiographic evaluation.

Patients will be identified for potential enrollment to the study by physician investigators at Robert Wood Johnson University Hospital (RWJUH), Robert Wood Johnson Somerset, University Orthopaedic Associates, and St. Peter's University Hospital Center for Ambulatory Resources (CARES). Once enrolled to the study, patients will be randomized to the two study arms in an alternating fashion. Every other patient will be randomized to one of the two groups. A potential source of bias exists in the fact that the surgeon will not be able to be entirely blinded to which group the patient is assigned, as the postoperative dressing is different between the two, so the surgeon must know which dressing to apply. Once assigned to a group preoperatively, patients will be counseled on their postoperative rehabilitation program. They will be given a pamphlet detailing restrictions, exercises, and motions allowed at each specific time point.

The patients will undergo distal radius open reduction and internal fixation utilizing a volar locking plate. Either a modified Henry volar approach or a trans-flexor carpi radialis (FCR) approach to the distal radius will be used. The specific type and brand of plate will be recorded. Immediate post-operative radiographs will be acquired. Patients assigned to the early mobilization group will be given a Velcro removable wrist splint to go home with, measured off their contralateral hand. All patients in both groups will be administered 10 Percocet pills (5 mg/325 mg) for postoperative pain. Patient consumption of pain medication will be captured at subsequent visits starting at 2 weeks.

For the early mobilization group, patients will be placed in a bulky soft dressing immediately after surgery. They will be made non-weight bearing, but active and passive motion of digits, forearm, elbow, and shoulder will be allowed with light functional tasks permitted as tolerated. Wrist motion within the soft dressing will be permitted as tolerated by patient. On postoperative day 3, patients will be advised to remove the dressing at home and begin home hand/wrist therapy. They will use a removeable Velcro wrist splint for nighttime wear and strenuous activity. This splint can be removed during normal activities of daily living (ADLs) and therapy. At this point, patients can shower without covering surgical site. However, soaking in standing water is not permitted. The first postoperative visit will be in 2 weeks. Sutures/staples will be removed if applicable. Patients will be advised to wean splint as tolerated with progressive weight bearing as pain permits. Patients will continue active and passive wrist motion exercises at home until 6 weeks post-op. From the 6-week timepoint onward, patients will have no restrictions. At the 6-week, 3 month, and 1 year postoperative visits, patients will have repeat radiographs taken, all measurements performed, and all questionnaires administered. All radiographs and visits for this study are standard of care. These data points are outlined below.

For the late mobilization group, immediately post-operatively patients will be placed in a plaster volar resting splint. They will be made non-weight bearing, with use of digits for light functional tasks permitted. They will be given home exercises for their fingers but will not yet resume wrist motion. At the first post-operative visit at the 2-week timepoint, the dressing and volar splint will be removed, along with sutures/staples if applicable. Patients will be converted to removeable Velcro wrist splint for nighttime and strenuous activity, which can be removed during normal ADLs and therapy. Patients will be given a list of home exercises to be performed as a pamphlet. Patients will be advised to wean splint as tolerated with progressive weight bearing as pain permitted. They will continue active and passive wrist motion exercises at home until 6 weeks post-op. From the 6-week timepoint onward, patients will have no restrictions. At the 6-week, 3 month, and 1 year postoperative visits, patients will have repeat radiographs taken, all measurements performed, and all questionnaires administered.

As stated, the follow-up visits for this study will be at 2 weeks, 6 weeks, 3 months, and 1 year. At each visit the patients will have radiographs taken, questionnaires administered, and quantitative testing done to assess range of motion and strength. Details further outlined below.

ELIGIBILITY:
Inclusion Criteria:

* DRF requiring volar plate fixation per physician investigator
* No medical comorbidities which would prevent them from having surgery per physician investigator
* Intra- or extra-articular DRF

Exclusion Criteria:

* Open fractures
* Comminuted fractures
* Polytrauma
* Bilateral DRFs
* Previous contralateral wrist injury that could limit comparison
* Additional ipsilateral fracture (except ulnar styloid - this will be recorded, but not an exclusion criteria)
* Pathologic fractures
* Additional fixation methods utilized (dorsal plate, K-wire, external fixator, etc.)
* Bone graft use
* Inability to comply with treatment protocol or follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Non-operative Hand Active Wrist Flexion | 6 weeks
  Wrist on the non-operated hand is flexed by subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Flexion | 3 months
  Wrist on the non-operated hand is flexed by subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Flexion | 1 year
  Wrist on the non-operated hand is flexed by subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Flexion | 6 weeks
  Wrist on the non-operated hand is flexed by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Flexion | 3 Months
  Wrist on the non-operated hand is flexed by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Flexion | 1 Year
  Wrist on the non-operated hand is flexed by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Extension | 6 weeks
  Wrist on the non-operated hand is extended by subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Extension | 3 Months
  Wrist on the non-operated hand is extended by subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Extension | 1 Year
  Wrist on the non-operated hand is extended by subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Extension | 6 weeks
  Wrist on the non-operated hand is extended by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Extension | 3 Months
  Wrist on the non-operated hand is extended by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Extension | 1 Year
  Wrist on the non-operated hand is extended by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Extension | 6 weeks
  Wrist on the operated hand is extended by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Extension | 3 Months
  Wrist on the operated hand is extended by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Extension | 1 Year
  Wrist on the operated hand is extended by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Extension | 6 weeks
  Wrist on the operated hand is extended by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Extension | 3 Months
  Wrist on the operated hand is extended by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Extension | 1 Year
  Wrist on the operated hand is extended by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Flexion | 6 weeks
  Wrist on the operated hand is flexed by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Flexion | 3 Months
  Wrist on the operated hand is flexed by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Flexion | 1 Year
  Wrist on the operated hand is flexed by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Flexion | 6 weeks
  Wrist on the operated hand is flexed by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Flexion | 3 Months
  Wrist on the operated hand is flexed by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Flexion | 1 Year
  Wrist on the operated hand is flexed by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Supination | 6 Weeks
  Wrist on the non-operated hand is actively supinated by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Supination | 3 Months
  Wrist on the non-operated hand is actively supinated by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Active Wrist Supination | 1 Year
  Wrist on the non-operated hand is actively supinated by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Supination | 6 Weeks
  Wrist on the non-operated hand is passively supinated by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Supination | 3 Months
  Wrist on the non-operated hand is passively supinated by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Non-operative Hand Passive Wrist Supination | 1 Year
  Wrist on the non-operated hand is passively supinated by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Supination | 6 Weeks
  Wrist on the operated hand is actively supinated by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Supination | 3 months
  Wrist on the operated hand is actively supinated by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Active Wrist Supination | 1 Year
  Wrist on the operated hand is actively supinated by the subject and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Supination | 6 Weeks
  Wrist on the operated hand is passive supinated by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Supination | 3 Months
  Wrist on the operated hand is passive supinated by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles
Operative Hand Passive Wrist Supination | 1 Year
  Wrist on the operated hand is passive supinated by the observer and joint angle is measured using a goniometer, a specialized protractor for measuring joint angles

SECONDARY OUTCOMES:
Radiographic evaluation of volar tilt | 2 weeks
  volar tilt of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of volar tilt | 6 weeks
  volar tilt of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of volar tilt | 3 Months
  volar tilt of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of volar tilt | 1 Year
  volar tilt of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial inclination | 2 Weeks
  Radial inclination of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial inclination | 6 Weeks
  Radial inclination of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial inclination | 3 Months
  Radial inclination of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial inclination | 1 Year
  Radial inclination of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial height | 2 Weeks
  Radial height of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial height | 6 Weeks
  Radial height of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial height | 3 Months
  Radial height of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of radial height | 1 Year
  Radial height of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of ulnar variance | 2 Weeks
  Ulnar variance of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of ulnar variance | 6 Weeks
  Ulnar variance of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of ulnar variance | 3 Months
  Ulnar variance of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of ulnar variance | 1 Year
  Ulnar variance of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of articular step off | 2 Weeks
  Articular step off of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of articular step off | 6 Weeks
  Articular step off of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of articular step off | 3 Months
  Articular step off of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of articular step off | 1 Year
  Articular step off of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of healing | 2 Weeks
  Fracture healing of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of healing | 6 Weeks
  Fracture healing of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of healing | 3 Months
  Fracture healing of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of healing | 1 year
  Fracture healing of the injured wrist will be measured using imaging processing software for radiographs.
Radiographic evaluation of fractured ulnar styloid | 2 Weeks
  Fracturing of the ulna styloid of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured ulnar styloid | 6 Weeks
  Fracturing of the ulna styloid of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured ulnar styloid | 3 Months
  Fracturing of the ulna styloid of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured ulnar styloid | 1 Year
  Fracturing of the ulna styloid of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured scapholunate interval | 2 Weeks
  Widening of the scapholunate interval of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured scapholunate interval | 6 Weeks
  Widening of the scapholunate interval of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured scapholunate interval | 3 Months
  Widening of the scapholunate interval of the injured wrist will be evaluated using imaging processing software for radiographs.
Radiographic evaluation of fractured scapholunate interval | 1 Year
  Widening of the scapholunate interval of the injured wrist will be evaluated using imaging processing software for radiographs.
Visual Analog Scale for Pain Level (VAS) | 2 Weeks
  Pain is described using a VAS that ranges from 0 to 10 where 0 is no pain and 10 is the worst pain.
Visual Analog Scale for Pain Level (VAS) | 6 Weeks
  Pain is described using a VAS that ranges from 0 to 10 where 0 is no pain and 10 is the worst pain.
Visual Analog Scale for Pain Level (VAS) | 3 Months
  Pain is described using a VAS that ranges from 0 to 10 where 0 is no pain and 10 is the worst pain.
Visual Analog Scale for Pain Level (VAS) | 1 Year
  Pain is described using a VAS that ranges from 0 to 10 where 0 is no pain and 10 is the worst pain.
pain medication use | 2 weeks
  Records if subject is still using pain medication.
pain medication use | 6 weeks
  Records if subject is still using pain medication.
pain medication use | 3 months
  Records if subject is still using pain medication.
pain medication use | 1 year
  Records if subject is still using pain medication.
length of sick leave from work | 6 weeks
  Records the date of return to work if subject has returned to work
length of sick leave from work | 3 months
  Records the date of return to work if subject has returned to work
length of sick leave from work | 1 year
  Records the date of return to work if subject has returned to work
complications | 2 weeks
  hardware loosening, malunion, non-union, delayed union, hardware failure, loss of reduction, refracture, nerve palsy, weakness, paresthesia, neuropathy, tendon rupture, adhesion, infection, wound dehiscence
complications | 6 weeks
  hardware loosening, malunion, non-union, delayed union, hardware failure, loss of reduction, refracture, nerve palsy, weakness, paresthesia, neuropathy, tendon rupture, adhesion, infection, wound dehiscence
complications | 3 months
  hardware loosening, malunion, non-union, delayed union, hardware failure, loss of reduction, refracture, nerve palsy, weakness, paresthesia, neuropathy, tendon rupture, adhesion, infection, wound dehiscence
complications | 1 year
  hardware loosening, malunion, non-union, delayed union, hardware failure, loss of reduction, refracture, nerve palsy, weakness, paresthesia, neuropathy, tendon rupture, adhesion, infection, wound dehiscence
Surgical Satisfaction Questionnaire (SSQ-8) | 6 weeks
  A series of questions answered using a Likert Scale from 0 - "Very Unsatisfied" to 4 - "Very Satisfied." The score ranges from 0 - 100 with higher scores indicating higher satisfaction.
Surgical Satisfaction Questionnaire (SSQ-8) | 3 months
  A series of questions answered using a Likert Scale from 0 - "Very Unsatisfied" to 4 - "Very Satisfied." The score ranges from 0 - 100 with higher scores indicating higher satisfaction.
Surgical Satisfaction Questionnaire (SSQ-8) | 1 year
  A series of questions answered using a Likert Scale from 0 - "Very Unsatisfied" to 4 - "Very Satisfied." The score ranges from 0 - 100 with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Varghese, MD, Study Director — Research Assistant
Locations (1):
- University Orthopedics Associates, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No